CLINICAL TRIAL: NCT02175602
Title: Effect of a Combination of Daclatasvir, Asunaprevir, and BMS-791325 on the Pharmacokinetics of Selective Serotonin Reuptake Inhibitors in Healthy Subjects
Brief Title: Study of Drug Combination on Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AI443-116
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — Escitalopram; Sertraline; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 2 (Experimental): Sertraline (50 milligrams each morning) day 1-7, DCV 3DAA FDC + 75 mg BMS-791325 twice daily days 13 to 22, DCV 3DAA FDC + 75 mg BMS-791325 twice daily + Sertraline (50 milligrams each morning) days 23-29
  Interventions: Drug: Sertraline; Drug: DCV 3DAA FDC; Drug: BMS-791325
- Cohort 1 (Experimental): Escitalopram (10 milligrams each morning) day 1-7, DCV 3DAA FDC + 75 mg BMS-791325 twice daily days 13 to 22, DCV 3DAA FDC + 75 mg BMS-791325 twice daily + Escitalopram (10 milligrams each morning) days 23-29
  Interventions: Drug: Escitalopram; Drug: DCV 3DAA FDC; Drug: BMS-791325

INTERVENTIONS:
Drug: Escitalopram — 10 milligrams administered each morning
  Other Names: Lexapro
  Arms: Cohort 1
Drug: Sertraline — 50 milligrams administered each morning
  Other Names: Zoloft
  Arms: Cohort 2
Drug: DCV 3DAA FDC — Fixed dose combination (daclatasvir [DCV] 30 milligrams, asunaprevir [ASV] 200 milligrams, and BMS-791325 75 milligrams) one tablet administered twice daily
Drug: BMS-791325 — 75 milligrams single-agent film coated oral tablet administered twice daily

SUMMARY:
The purpose of this study is to assess the effect of Daclatasvir, Asunaprevir, and BMS-791325 on the pharmacokinetics of selective serotonin reuptake inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form

   a) Signed written informed consent must be obtained from the subjects in accordance with requirements of the study center's IRB or IEC before the initiation of any protocol-required procedures.
2. Target Population

   a) Healthy subjects as determined by no clinically significant deviation from normal in medical history, psychiatric history, physical examination findings, vital sign measurements, 12-lead ECG measurements, physical measurements, and clinical laboratory test results.
3. Age and Reproductive Status

   1. Males and females, ages 25 to 55 years, inclusive.
   2. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
   3. Women must not be breastfeeding.

Exclusion Criteria:

1. Any significant acute or chronic medical illness.
2. Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug (appendectomies with no complications are allowed at the investigator's discretion).
3. Any major surgery within 4 weeks of study drug administration.
4. Smokers (those who currently smoke, as well as those who have stopped smoking less than 6 months prior to the start of study drug administration).
5. Any other sound medical, psychiatric, and/or social reason as determined by the investigator.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Serial blood samples for plasma SSRI (selective serotonin reuptake inhibitor) of escitalopram or sertraline | Before dosing (0 hour) through 24 hours after SSRI administration on day 7 and day 29
Serial blood samples for determination of plasma concentrations of DCV (daclatasvir), ASV (asunaprevir), BMS-791325, and the metabolite BMS-794712 | Before dosing (0 hour) through 12 hours after SSRI administration on day 22 and day 29

SECONDARY OUTCOMES:
Safety assessments based on review of adverse events, vital sign measurements, electrocardiograms, physical examinations, and clinical laboratory tests. | Two to three months

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna Ogbaa, MD, Principal Investigator — PPD Development, LP